CLINICAL TRIAL: NCT05671783
Title: Different Types of Intraoperative Hypotension and Their Association With Post-anesthesia Care Unit Recovery
Brief Title: Intraoperative Hypotension and Post-anesthesia Care Unit Recovery
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-08/10
Record Dates: First submitted 2022-12-21; First posted 2023-01-05 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Post-induction Hypotension; Post Anesthesia Recovery; Hypotension; Intraoperative Hypotension
Keywords: Complication; Intraoperative Hypotension; PACU outcomes; PACU recovery; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-induction hypotension: Post-induction hypotension (pIOH) is a decrease during the first 20 min after anesthesia induction
  Interventions: Other: Hemodynamic observation of the patients.
- Maintenance intraoperative hypotension: maintenance intraoperative hypotension (mIOH) when there is a decrease of blood pressure 20th min after induction, with or without pIOH
  Interventions: Other: Hemodynamic observation of the patients.
- Normotensive patients: Patients with normotension during surgery.
  Interventions: Other: Hemodynamic observation of the patients.

INTERVENTIONS:
Other: Hemodynamic observation of the patients. — For the purposes of this study, we defined intraoperative hypotension as a decrease in mean blood pressure of 30% from baseline for a minimum of 5 minutes, including induction and maintenance of anesthesia. The measuring blood pressure method (noninvasive or invasive) depended on the surgical intervention's invasiveness and the patient's cardiac performance.
  As soon as the patients entered the PACU, the responsible nurses started the standard monitoring. Anesthesiologists constantly oversee all actions based on the patient's condition. Clinical observation for respiratory and gastrointestinal problems and all disorders were monitored. When in room air SO2 was <94, we started oxygen treatment with a 4 liter/minute nasal cannula, and in cases of nausea antiemetic was administered. The Modified Aldrete Score was used to discharge the patent.
  Other Names: Postoperative clinical observation

SUMMARY:
The underlying causative mechanism that leads to intraoperative hypotension (IOH) may vary depending on the stage of anesthesia and surgery, which determines different IOH types. Naturally, the incidence and severity of IOH types will differ, as will the incidence and severity of postoperative complications.

DETAILED DESCRIPTION:
Background The underlying causative mechanism that leads to intraoperative hypotension (IOH) may vary depending on the stage of anesthesia and surgery, which determines different IOH types. Naturally, the incidence and severity of IOH types will differ, as will the incidence and severity of postoperative complications.

Methods The investigators conducted a data-based observational study that included 4776 patients. Post-induction hypotension (pIOH) is defined as a decrease during the first 20 min after anesthesia induction and maintenance intraoperative hypotension (mIOH) when there is a decrease of blood pressure 20th min after induction, with or without pIOH.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Underwent elective surgery
* Received general anesthesia
* Planned overnight stay in the hospital after surgery

Exclusion Criteria:

* Under 18 years of age
* Cardiac surgery
* Transplant surgery
* Preoperatively receiving vasoactive drugs
* Patients with mechanical circulatory support
* Pediatric surgery
* Patients from ICU
* Patients with scheduled postoperative ICU admissions

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We conducted a data-based observational study. Only routinely documented patient data was considered in the recent study. All patients' preoperative and postoperative recovery room data is recorded in a virtual environment. Data describing consecutive patients were collected until the patient was discharged to a ward. Data included demographics, comorbidities, perioperative hemodynamic parameters, duration of PACU, complications in PACU, and non-planned intensive care admission.
Sampling Method: Probability Sample
Enrollment: 4776 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Effect of IOH types on PACU recovery (Duration) | From the preoperative first monitorization of the patient in the operating room until until discharege from the PACU (0-720 minutes).
  The underlying causative mechanism that leads to IOH may vary depending on the stage of anesthesia and surgery, which determines different IOH types; therefore recovery after them will differ.
  care unit (PACU) recovery, especially duration and complications in the PACU.

SECONDARY OUTCOMES:
PACU recovery | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Compare the effect of intraoperative hypotension types on PACU recovery to the effect of other factors influencing PACU recovery.

OTHER OUTCOMES:
Effect of IOH types on PACU duration | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Different IOH types may have a different impact on the PACU duration.
Effect of IOH types on PACU complications | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Different IOH types have a different impact on the PACU's complication rate.
Intraoperative hypotension | From the preoperative first monitorization of the patient in the operating room until extubation and transfer to the PACU (0-480 minutes).
  Decrease in mean blood pressure of 30% from baseline for a minimum of 5 minutes, including induction and maintenance of anesthesia.
pIOH | From the preoperative first monitorization of the patient in the operating room to the 20th minute after anesthesia induction.
  Decrease in mean blood pressure of 30% from baseline during the first 20 min after anesthesia induction.
mIOH | From the 20th minute after anesthesia induction until extubation and transfer to the PACU (between 20- 480 minutes).
  Decrease of blood pressure 20th min after induction, with or without pIOH.
PACU complications: desaturation | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Postoperative SpO2<%90
PACU complications: Arrhythmia | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Irregular heartbeat
PACU complications: Bradycardia | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Postoperative heart rate < 40 min
PACU complications: Tachycardia | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Postoperative heart rate >100 min >100 min-1 Heart rate >100 min-1
PACU complications: Gastrointestinal complications | Postoperatively from the patient's arrival to the PACU until discharge (0-240 minutes).
  Include nausea and vomiting
Unplanned ICU admission | From the preoperative first monitorization of the patient in the operating room until until discharege from the PACU (0-720 minutes).
  When ICU bed reservation is not considered in the preoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Lerzan Dogan, MD, Study Chair — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data on patients is available.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: valid reason

REFERENCES:
- [Background] Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007 Aug;107(2):213-20. doi: 10.1097/01.anes.0000270724.40897.8e. PMID 17667564
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Background] Gregory A, Stapelfeldt WH, Khanna AK, Smischney NJ, Boero IJ, Chen Q, Stevens M, Shaw AD. Intraoperative Hypotension Is Associated With Adverse Clinical Outcomes After Noncardiac Surgery. Anesth Analg. 2021 Jun 1;132(6):1654-1665. doi: 10.1213/ANE.0000000000005250. PMID 33177322
- [Background] Waddle JP, Evers AS, Piccirillo JF. Postanesthesia care unit length of stay: quantifying and assessing dependent factors. Anesth Analg. 1998 Sep;87(3):628-33. doi: 10.1097/00000539-199809000-00026. PMID 9728843
- [Background] Chen B, Pang QY, An R, Liu HL. A systematic review of risk factors for postinduction hypotension in surgical patients undergoing general anesthesia. Eur Rev Med Pharmacol Sci. 2021 Nov;25(22):7044-7050. doi: 10.26355/eurrev_202111_27255. PMID 34859868
- [Background] Jor O, Maca J, Koutna J, Gemrotova M, Vymazal T, Litschmannova M, Sevcik P, Reimer P, Mikulova V, Trlicova M, Cerny V. Hypotension after induction of general anesthesia: occurrence, risk factors, and therapy. A prospective multicentre observational study. J Anesth. 2018 Oct;32(5):673-680. doi: 10.1007/s00540-018-2532-6. Epub 2018 Jul 19. PMID 30027443
- [Derived] Dogan L, Yildirim SA, Sarikaya T, Ulugol H, Gucyetmez B, Toraman F. Different Types of Intraoperative Hypotension and their Association with Post-Anesthesia Care Unit Recovery. Glob Heart. 2023 Aug 11;18(1):44. doi: 10.5334/gh.1257. eCollection 2023. PMID 37577293